CLINICAL TRIAL: NCT04598243
Title: Treatment of Fibromyalgia and CFS With Ribose, Ashwagandha, Rhodiola, Licorice, Schisandra and Green Tea Extract
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Practitioners Alliance Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAN-SES 1-2020
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Fibromyalgia; CFS
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of CFS/FMS with the nutritional combination (Experimental)
  Interventions: Dietary Supplement: Smart Energy System

INTERVENTIONS:
Dietary Supplement: Smart Energy System — A nutritional /herbal combination

SUMMARY:
Is a combination of Ribose, Ashwagandha, Rhodiola, Schisandra, licorice, and green tea extract helpful in CFS and FIbromyalgia?

DETAILED DESCRIPTION:
Ribose has been shown to be very helpful in CFS and fibromyalgia. Many studies have also shown benefit for the symptoms of these conditions from Ashwagandha, Rhodiola, Schisandra, licorice, and green tea extract. The study is undertaken as an early open label study to check for the efficacy of a proprietary combination of these

ELIGIBILITY:
Inclusion Criteria:

1. be diagnosed with CFS and/or fibromyalgia
2. live in the United States 3 - be over 18 years of age

Exclusion Criteria:

1. pregnancy
2. Diabetes
3. Hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-07-04 (Estimated); Study Completion 2021-07-04 (Estimated)

PRIMARY OUTCOMES:
VAS | 4-6 weeks
  A composite VAS of Fatigue, Pain, Sleep, Cognition and overall well-being. These are each on a 1-10 scale with the same units, with 10 being healthy. The composite sum total of all of these (0-50) will be used as a single outcome measure

CONTACTS AND LOCATIONS:
Locations (1):
- Kona Research Center, Kailua, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No